CLINICAL TRIAL: NCT01822262
Title: All the Phases Study Will be Operated by the Department of Hepatobiliary Surgery, The Affiliated Hospital of Guiyang Medical College
Brief Title: Contrastive Study for Minimally Invasive Cholecystolithotomy With Gallbladder Reservation and Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengyi Sun (Other)
Responsible Party: Sponsor-Investigator, Chengyi Sun, Department of Hepatobiliary Surgery, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GYGDWK-01
Record Dates: First submitted 2013-03-14; First posted 2013-04-02 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2016-03

CONDITIONS: Gallstones
Keywords: Cholecystolithotomy with gallbladder reservation; cholecystolithiasis
MeSH Terms: conditions — Gallstones; Cholecystolithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gallbladder reservation (Experimental): Patients in trial group all took minimally invasive cholecystolithotomy with gallbladder reservation
  Interventions: Procedure: minimally invasive cholecystolithotomy with gallbladder reservation
- laparoscopiccholecystectomy (Experimental): Patients in control group all received LC.
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: minimally invasive cholecystolithotomy with gallbladder reservation
  Arms: gallbladder reservation
Procedure: laparoscopic cholecystectomy
  Other Names: LC
  Arms: laparoscopiccholecystectomy

SUMMARY:
To explore the therapeutic effects for treatment of cholecystolithiasis by minimally invasive cholecystolithotomy with gallbladder reservation and laparoscopic cholecystectomy. Method： patients with cholecystolithiasis who received minimally invasive Cholecystolithotomy with gallbladder reservation and patients with cholecystolithiasis who received laparoscopic cholecystectomy(LC) in The Affiliated Hospital of Guiyang Medical College from May 2011 to December 2013. Patients who received minimally invasive cholecystolithotomy with gallbladder reservation as trial group, patients who received LC as control group.the overall follow-up period is 1 year. Then the investigators statistically analyze improvement of cholecystolithiasis symptoms in every group, thickness of gall bladder wall, the gallbladder function and the rate of the recurrence of cholesterol gallstone in trial group.

DETAILED DESCRIPTION:
The investigators Prospect： Minimally invasive cholecystolithotomy with gallbladder reservation is meaningful for recovering the function of gallbladder.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of calculous cholecystitis.

Exclusion Criteria:

* Gallbladder's wall >3mm, atrophied gallbladder,gallstone obstruct the Hartmann's pouch.
* Abdominal ultrasound display the contractibility of gallbladder is poor.
* The aged patients with bad heart and lung function.
* Patients who has acute cholecystitis,pancreatitis,pancreaticobiliary diseases, especially choledocholithiasis.
* Pregnant or lactational women.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The contraction function of the gallbladder | Participants will be followed for overall 1 year after surgery
  Measure the participants' contraction function of gallbladder by the trial for contraction function of gallbladder

SECONDARY OUTCOMES:
The thickness of gallbladder wall | Participants will be followed for overall 1 year after surgery
  Measure the participants' thickness of gallbladder wall by abdominal ultrasonography after surgery

OTHER OUTCOMES:
The improvement of cholelith symptoms | Participants will be followed for overall 1 year after surgery
The recurrence rate of gallstone | Participants will be followed for overall 1 year after surgery
  Measure the participants' recurrence rate of gallstone by abdominal ultrasonography after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chengyi Sun, M.D, Study Chair — The Affiliated Hospital of Guiyang Medical College
Locations (1):
- The Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou, China